CLINICAL TRIAL: NCT03798522
Title: Analgesic Efficacy of Erector Spinae Plane Block Versus Opioid Based General Anesthesia During Laparoscopic Bariatric Surgery; a Randomized Controlled Study
Brief Title: Erector Spinae Plane Block Versus Opioid Based General Anesthesia During Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohammed El-Hadi Shoukat Mohammed, lecturer of anesthesia, pain management and surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N-42-2018
Record Dates: First submitted 2018-12-27; First posted 2019-01-10 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Bariatric Surgery Candidate; Morbid Obesity; Visceral Pain
Keywords: ultrasound guided regional blocks; laparoscopic surgery; erector spinae plane block
MeSH Terms: conditions — Obesity, Morbid; Visceral Pain | interventions — Nalbuphine

STUDY DESIGN:
Intervention Model Description: * erector spinae plane block group (ESPB)
  * general anesthesia group (GA)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erector spinae plane block group (ESPB) n=14 (Experimental): Bilateral ultrasound guided erector spinae plane block will be performed in the lateral position at T7 vertebrae and before induction of GA. 20 ml of local anesthetic solution (20 ml bupivacaine (Sunnypivacaine, Sunny pharmaceutical, Egypt) 0.25%) will be injected in-plane into the ESP. This procedure will be repeated on the other side taking care not to exceed the maximum recommended doses (2 mg/kg of IBW for bupivacaine) and then GA will be conducted .
  Interventions: Procedure: bilateral ultrasound guided erector spinae plane block
- general anesthesia group (GA) n= 14 (Active Comparator): these patients will receive iv nalbuphine in dose of 2mg /kg according to ideal body weight after induction of GA
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Procedure: bilateral ultrasound guided erector spinae plane block — ESPB on both sides at T7 before GA
  Other Names: ESPB
  Arms: erector spinae plane block group (ESPB) n=14
Drug: Nalbuphine — in nalbuphine for analgesia after GA
  Other Names: GA
  Arms: general anesthesia group (GA) n= 14

SUMMARY:
bilateral continuous erector spinae plane blockade may represent a valuable alternatives to thoracіc epidurals analgaesіa in treatment of thoracic neuropathic pain.

There were 3 cases reported in 2017 suggested that the erector spinae plane block provides visceral abdominal analgesia in bariatric surgery and at end of the report they recommended further clinical investigation. The investigators hypothesіzed that performing the erector spinae plane (ESP) block at T7 would provide effective abdominal analgaesіa іn patients undergone laparoscopic bariatric surgery. The investigators aimed to compare the analgesic effect of erector spinae plane block and opioid based general anesthesia for laparoscopic bariatric surgeries.

DETAILED DESCRIPTION:
The investigators hypothesized that, erector spinae plane block will provide good analgesia for patients undergoing laparoscopic bariatric surgery with less complication compared to opioid based general anesthesia. The visual analogue scale (VAS) will be explained clearly to all participants before conduction of anesthesia. All the drugs will be calculated according to the ideal body weight (IBW).A low-frequency (2-5 MHz) curved array ultrasound probe (Mindray®, China) will be used. In the 1st group: bilateral ultrasound-guided erector spinae plane block will be performed under complete aseptic conditions in the lateral position at T7 vertebrae and before induction of general anesthesia. An 8-cm echogenic 22-G block needle will be inserted in-plane. A total of 20 ml of local anesthetic solution (20 ml bupivacaine (Sunnypivacaine, Sunny pharmaceutical, Egypt) 0.25%) will then be injected into the erector spinae plane. This procedure will be repeated on the contralateral side taking care not to exceed the maximum recommended doses (2 mg/kg of IBW for bupivacaine). In the 2nd group: the investigator will give intravenous nalbuphine in a dose of 2mg /kg according to ideal body weight after induction of general anesthesia. All participants will be given 1 gram of intravenous paracetamol (15 mg/Kg), together with 4 mg ondansetron 10 min prior to the end of surgery for postoperative nausea and vomiting prophylaxis.

Intraoperatively, any increase in heart rate and/or arterial blood pressure 10 min after intubation by more than 20% of baseline values in response to surgical stimulus or thereafter throughout the whole operation will be managed by intravenous administration of fentanyl 0.5 µg/Kg. VAS score will be assessed 30 min after extubation and when the VAS score exceeded 4/10, rescue analgesia in the form of IV nalbuphine 5 mg will be administered. Another dose of rescue analgesia can be given in the post anesthesia care unit (PACU) if the VAS still more than 4 after 60 min of extubation. If still high, Ketorolac 60 mg will be given by intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18 <60
* Obese patients 40˂ Body mass index(BMI) ˂50
* Both sexes
* American Society of Anesthesiologists(ASA) physical status classes II and III
* Patients scheduled for laparoscopic bariatric surgery i.e. sleeve gastrectomy and/or Roux-en-Y gastric bypass (RYGB)surgeries

Exclusion Criteria:

* Refusal of regional block
* Patients with neurological, psychological disorders or those lacking cooperation
* Patients scheduled for concomitant laparoscopic cholecystectomy or paraumbilical hernia repair or those with history of previous bariatric surgery or obstructive sleep apnea
* Patients with anatomic abnormalities at site of injection, skin lesions or wounds at site of proposed needle insertion.
* Patients with bleeding disorders defined as (INR >2) and/ or (platelet count <100,000/µL)
* Patients with hepatic disease e.g. liver cell failure or hepatic malignancy or hepatic enlargement.
* Patients who are allergic to amide local anesthetics.
* Cases converted to open surgery will also be excluded from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The duration of analgesic effect in minutes | defined as the time n minutes between finishing the block technique in ESPB group or after administration of nalbuphine in GA-group, and the request of first dose of postoperative analgesics) when VAS is more than 4 during the 1st 8 hours postoperatively
  The duration of analgesic effect is indicated by the 1st analgesic requisite after measurement of VAS

SECONDARY OUTCOMES:
mean arterial blood pressure changes | intraoperative and post extubation in the 1st hour
  mean arterial blood pressure will be assessed and measured in mmHg non invasively
Nalbuphine consumption | total dose given post operatively up to 1 hour postoperatively
  in mg
visual analogue scale (VAS) for assessment of postoperative pain | at 30 minutes, 45 minutes and 60 minutes, 4 hours and 8 hours after surgery
  in numbers, normal scale ranges from 0 to 10 with 0 means no pain and 10 means worst pain imaginable. if VAS score exceeded 4/10; this will be considered insufficient analgesia and participant will be given rescue analgesia
Block failure rate | in the first hour postoperatively
  patient required more than two 5mg doses of nalbuphine
Resumption of peristalsis | postoperatively up to 48 hours postoperatively
  in hours
incidence of adverse effects | postoperative up to 48 hours
  postoperative nausea and vomiting, urinary retention, hematoma formation, local anesthetic toxicity and need of postoperative ICU or mechanical ventilation
Incidence of shoulder pain | postoperativey up to 24 hours
  percent
length of hospital stay | postoperative up to 28 days postoperatively
  in days
heart rate | intraoperatively and throughout one hour postextubation
  heart rate in beat per minute will be measured
Failure rate of the ESP block | in the first hour postoperatively
  the block will be considered a failed block if the patient required more than two 5mg doses of nalbuphine

OTHER OUTCOMES:
demographic data | during 30 minutes preoperatively
  age, sex, ASA class, co-morbidities
duration of surgery | from skin incision up to skin closure
  in minutes
weight | during 30 minutes preoperatively
  kilograms
height | during 30 minutes preoperatively
  meter
body mass index (BMI) | uring 30 minutes preoperatively
  weight in kilograms divided by square height in meter

CONTACTS AND LOCATIONS:
Locations (1):
- Hany Mohammed El-Hadi Shoukat Mohammed, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
yes
Supporting Information: Study Protocol, SAP
Time Frame: 9 months
Access Criteria: Researchgate.gov